CLINICAL TRIAL: NCT01511523
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Effect of RGMA001 on Patients With Non Alcoholic Fatty Liver Disease (NAFLD).
Brief Title: Study to Evaluate the Effect of RGMA001 on Patients With Non Alcoholic Fatty Liver Disease (NAFLD)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Biovil Research Group, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: BVL-001
Record Dates: First submitted 2012-01-13; First posted 2012-01-18 (Estimated); Last update posted 2012-03-16 (Estimated); Status verified 2012-01

CONDITIONS: Non Alcoholic Fatty Liver Disease
Keywords: Liver; Fatty; Non Alcoholic; Vitamin E; Silymarin; Carnitine; Supplement; NAFLD
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- RGMA001 (Active Comparator): Proprietary blend of Vitamin E, Silymarin, and Carnitine.
  Interventions: Dietary Supplement: RGMA001
- Sugar Pill (Placebo Comparator): No treatment.
  Interventions: Dietary Supplement: Sugar Pill

INTERVENTIONS:
Dietary Supplement: RGMA001 — 3 capsules administered BID once a day.
  Arms: RGMA001
Dietary Supplement: Sugar Pill — Placebo
  Arms: Sugar Pill

SUMMARY:
A research study of a compound containing vitamin E, silymarin and carnitine, three over the counter supplements. The investigators hope to learn if the new supplement can safely and successfully treat fatty liver disease or Non Alcoholic Fatty Liver Disease (NAFLD).

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients age 18 years and older.
2. A clinical or histologic or radiographic diagnosis of NAFLD.
3. Abnormities above normal range in hepatic function testing consisting of panels containing ALT, AST, AP, Total bilirubin and albumin.
4. Negative urine pregnancy test (for females of childbearing potential) collected at screening followed by another negative serum pregnancy test collected within 24 hours prior to the first dose of study drug.
5. Female patients of childbearing potential must be on adequate birth control.
6. Willingness to give written informed consent and willingness to participate in and comply with the study requirements.

Exclusion Criteria:

1. History of having received any investigational drug ≤ 3 months prior to the first dose of study drug or the expectation that such drugs will be used during the study. Patients enrolled in this study cannot be enrolled in another study for either research, diagnostic or treatment purposes.
2. Positive test at screening for anti-HAV IgM Ab, HBsAg, anti-HBc IgM Ab, or anti-HIV Ab.
3. History or other evidence of a medical condition associated with chronic liver disease other than NAFLD (e.g., hemochromatosis, viral or autoimmune hepatitis, Wilson's disease, α1-antitrypsin deficiency, alcoholic liver disease, and/or toxin exposure).
4. Females who are pregnant or breast feeding.
5. Platelet count < 90 x 103 / µL (< 90 x 109 /L) at screening.
6. Hemoglobin (Hgb) concentration < 12 g/dL (< 120 g/L) in females or < 13 g/dL (< 30 g/L) in males at screening.
7. Any patient with a baseline increased risk for anemia (e.g., thalassemia, sickle cell anemia, spherocytosis, history of gastrointestinal bleeding) or for whom anemia would be medically problematic.
8. Patients with history of severe psychiatric disease, including psychosis and/or severe depression, characterized by a suicide attempt, hospitalization for psychiatric disease, or a period of disability as a result of psychiatric disease must have a psychiatric evaluation at screening to ensure the patient is now stable and the patient must agree to have continued monitoring by a mental health specialist at least every 4 weeks during the study.
9. History of immunologically mediated disease [(e.g., vasculitis, cryoglobulinemia, inflammatory bowel disease, idiopathic thrombocytopenic purpura, lupus erythematosus, autoimmune hemolytic anemia, scleroderma, severe psoriasis (defined as affecting > 10% of the body, where the palm of one hand equals 1%, or if the hands and feet are affected), rheumatoid arthritis requiring more than intermittent nonsteroidal anti-inflammatory medications for management, etc.
10. Patients with evidence of decompensated liver disease including but not limited to ascites, esophageal varices, and hepatic encephalopathy.
11. History of any systemic anti-neoplastic or immunomodulatory treatment (including supraphysiologic doses of steroids and radiation) 6 months prior to the first dose of study drug or the expectation that such treatment will be needed at any time during the study
12. History or other evidence of decompensated liver disease or Child-Pugh Grade B or higher [Appendix 1], coagulopathy, hyperbilirubinemia, hepatic encephalopathy, hypoalbuminemia, ascites, and bleeding from esophageal varices are conditions consistent with decompensated liver disease.
13. One or more of the following conditions: (1) poorly controlled hypertension, OR (2) screening or baseline blood pressure ≥ 160 mmHg for systolic OR (3) screening or baseline blood pressure ≥ 100 mmHg for diastolic blood pressure.
14. History of bleeding disorders or anticoagulant use
15. Type I or II diabetes with HbA1C > 8.5% at screening.
16. History or other evidence of chronic pulmonary disease associated with functional limitation.
17. History of severe cardiac disease (e.g. NYHA Functional Class III or IV, myocardial infarction within 6 months, ventricular tachyarrhythmias requiring ongoing treatment, unstable angina or other significant cardiovascular disease). Patients with stable coronary artery disease (e.g., 6 months after by-pass surgery, angioplasty with or without stent placement, etc.) as confirmed by a cardiologist will be permitted. In addition, patients with documented or presumed unstable coronary artery disease, stable or unstable cardiovascular disease or cerebrovascular disease, or second or third degree heart block should not be enrolled.
18. History of uncontrolled severe seizure disorder.
19. Evidence of an active or suspected cancer, or a history of malignancy within the last 2 years, with the exception of patients with basal cell carcinoma that has been excised and cured.
20. Poorly controlled thyroid dysfunction.
21. History or other evidence of a clinically relevant ophthalmologic disorder due to diabetes mellitus or hypertension or history or other evidence of severe retinopathy (e.g., cytomegalovirus, macular degeneration).
22. History of major organ transplantation with an existing functional graft.
23. History or other evidence of severe illness, or any other conditions which would make the patient, in the opinion of the investigator, unsuitable for the study.
24. Any herbal supplements containing silymarin, tocopherol, vitamin C, bioflavins, curcumin. For complete list see appendix.3
25. Consumption of any nutrients know to possess antioxidant activity
26. Evidence of excessive alcohol, drug or substance abuse (excluding marijuana use) within 1 year of first dose.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-01; Primary Completion 2012-10 (Estimated); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
Efficacy | 30 weeks
  Normalization of hepatic AST, ALT, y-GT, albumin, alkaline phosphatase and total bilirubin.

SECONDARY OUTCOMES:
Safety | 30 weeks
  Vital signs, BMI, symptom directed physical exam, pregnancy tests, laboratory tests (hematology, and chemistry), clinical adverse events, dose modifications and treatment discontinuations related to adverse events or laboratory abnormalities.

CONTACTS AND LOCATIONS:
Overall Officials: John Poulos, MD, Principal Investigator — Cumberland Research Associates
Locations (1):
- Cumberland Research Associates, LLC, Fayetteville, North Carolina, United States